CLINICAL TRIAL: NCT02207361
Title: A Randomized Prospective Clinical Trial of Paclitaxel in Combination With Carboplatin Versus Paclitaxel Plus Epirubicin as First-Line Treatment in Metastatic Breast Cancer
Brief Title: Paclitaxel in Combination With Carboplatin Versus Paclitaxel Plus Epirubicin in Metastatic Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIH-TZS-20140421-02
Record Dates: First submitted 2014-04-22; First posted 2014-08-04 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2013-06

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — CP protocol; Paclitaxel; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel, Carboplatin，injection (Experimental): Paclitaxel: 175mg/m2, IV, d1 Carboplatin: AUC 5, IV, d1 Every 21 days to 1 course of treatment.
  Interventions: Drug: Paclitaxel, Carboplatin
- Paclitaxel, Epirubicin，injection (Active Comparator): Paclitaxel: 175mg/m2, IV, d1 Epirubicin: 60-80mg/m2, IV, d1 Every 21 days to 1 course of treatment.
  Interventions: Drug: Paclitaxel, Epirubicin

INTERVENTIONS:
Drug: Paclitaxel, Carboplatin — Paclitaxel: 175mg/m2, IV, d1 Carboplatin: AUC 5, IV, d1 Every 21 days to 1 course of treatment.
  Arms: Paclitaxel, Carboplatin，injection
Drug: Paclitaxel, Epirubicin — Paclitaxel: 175mg/m2, IV, d1 Epirubicin: 60-80mg/m2, IV, d1 Every 21 days to 1 course of treatment.
  Arms: Paclitaxel, Epirubicin，injection

SUMMARY:
Paclitaxel plus Epirubicin in metastatic breast cancer is a recommended scheme in National Comprehensive Cancer Network (NCCN) guideline. Paclitaxel in Combination with Carboplatin is also effective in Metastatic Breast Cancer (MBC) in some clinical study with small sample.

DETAILED DESCRIPTION:
A Randomized Prospective Clinical Trial of Paclitaxel in Combination with Carboplatin Versus Paclitaxel plus Epirubicin as First-Line Treatment in Metastatic Breast Cancer. The primary endpoints of the study is progression free survival (PFS). The secondary endpoints are overall response rate (ORR), overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

* female ≥ 18 years old, ECOG 0-2 or KPS≥60, Expected lifetime more than 12 weeks.

Exclusion Criteria:

* Pregnancy, Paclitaxel, platinum and anthracycline-based drugs' allergy, Severe Infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
RECIST 1.1 | -7 days

CONTACTS AND LOCATIONS:
Overall Officials: Zhongsheng Tong, Master, Study Director — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Egger SJ, Chan MMK, Luo Q, Wilcken N. Platinum-containing regimens for triple-negative metastatic breast cancer. Cochrane Database Syst Rev. 2020 Oct 21;10(10):CD013750. doi: 10.1002/14651858.CD013750. PMID 33084020